CLINICAL TRIAL: NCT04290793
Title: Pyrotinib Combined With Epirubicin and Cyclophosphamide Followed by Docetaxel Plus Trastuzumab in Neoadjuvant Therapy of HER2-positive Early Breast Cancer: a Single-arm, Open-label, Multicenter Phase II Clinical Trial
Brief Title: Neoadjuvant Chemotherapy With Pyrotinib, Epirubicin and Cyclophosphamide Followed by Taxanes and Trastuzumab for HER-2+ Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Liu Yunjiang, Director, Hebei Medical University Fourth Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRHB-CB001
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Epirubicin; Cyclophosphamide; Taxoids; Trastuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Active Comparator): Patients will receive the test drug (Pyrotinib) combined with Epirubicin and Cyclophosphamide followed by Taxanes and Trastuzumab with Pyrotinib
  Interventions: Drug: Pyrotinib; Drug: Epirubicin; Drug: Cyclophosphamide; Drug: Taxanes; Biological: Trastuzumab

INTERVENTIONS:
Drug: Pyrotinib — 400mg administered as continuous oral once daily from the first day of the study
Drug: Epirubicin — 90mg/m^2 d1 iv Q2W for 4 cycles
Drug: Cyclophosphamide — 600 mg/m^2 d1 iv Q2W for 4 cycles
Drug: Taxanes — Albumin paclitaxel（125mg/m2 d1、8 iv Q3W for 4 Cycles）/Docetaxel(100mg/m2 d1 iv Q3W for 4 Cycles )
Biological: Trastuzumab — the first cycle is a loading dose of 8 mg / kg, followed by 6 mg / kg. Iv Q3W

SUMMARY:
This is a prospective, open label, single-arm study to evaluate the efficacy and safety of neoadjuvant pyrotinib in HER2+ breast cancer patients

ELIGIBILITY:
Inclusion Criteria:

1. Female breast cancer patients at the age of >= 18 years and <= 70 years who received first treatment；
2. Pathologically confirmed HER2-positive invasive breast cancer（which is defined as the immunohistochemistry score of > 10% immunoreactive cells being 3+ or in situ hybridization results showing HER2 gene amplification），regardless of hormone receptor status (ER and PR)；
3. According to the 2019 CSCO BC guidelines: When HER-2 positive is used as the standard for preoperative neoadjuvant therapy for breast cancer, the tumor is larger than 2 cm；
4. The Eastern Tumor Collaborative Group (ECOG) has a physical status score of ≤1；
5. The functional level of the main organs must meet the following requirements ： 1) blood routine test: hemoglobin (Hb) ≥ 90g/L;Neutrophils (ANC) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 90 × 10^9/L; 2) Blood biochemistry: Total bilirubin (TBIL) ≤ 1.5 upper limit of normal value (ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 1.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; Urea nitrogen (BUN) and creatinine (Cr) ≤ 1.5 × ULN; 3) Heart color ultrasound: Left ventricular ejection fraction (LVEF) ≥ 55%;
6. Women of childbearing age, tested negative for serum pregnancy test 7 days before randomization，and willing to use appropriate methods during the trial and within 8 weeks after the last administration of the test drug;
7. A volunteer to participate in the study; provision of written informed consent; good compliance and willing to cooperate during the follow-up.

Exclusion Criteria:

1. Known history of hypersensitivity to pyrotinib or any of it components;
2. Patients have previously received antitumor treatment or radiation therapy for any malignant tumor (except for cervical carcinoma in situ and basal cell carcinoma that have been cured);
3. Patients underwent major breast cancer-free surgery within 4 weeks and have not fully recovered;
4. Subjects that are unable to swallow tablets,intestinal obstruction or dysfunction of gastrointestinal absorption;
5. Patients with severe heart disease or discomfort who cannot be treated;
6. The patient suffers from mental illness or psychotropic substance abuse and cannot cooperate;
7. Pregnant or lactating women;
8. Less than 4 weeks from the last clinical trial;
9. Patients participating in other clinical trials at the same time
10. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
tpCR | immediately after surgery
  It is defined as the absence of residual invasive carcinoma in the resected breast cancer specimens stained with hematoxylin and eosin, and no cancer metastasis in all ipsilateral lymph node samples, after completion of neoadjuvant therapy and surgery.

SECONDARY OUTCOMES:
Objective Response Rate(ORR) | 2 years
  Baseline to measured stable disease
Disease-free survival(DFS) Baseline to measured date of recurrence or death from any cause | 3 years
  Baseline to measured date of recurrence or death from any cause
bpCR | immediately after surgery
  After neoadjuvant chemotherapy and surgery, breast was free of any invasive cancer
Adverse Events rate | 1-year
  Evaluate the nature, incidence and severity of chemotherapy adverse events according to CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China